CLINICAL TRIAL: NCT05262049
Title: Comparison of Intermittent Compression-decompression With Glides and Conventional Physical Therapy Protocol for Knee Osteoarthritis
Brief Title: Comparison of Intermittent Compression-decompression With Glides for Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Riphah/RCRS/REC/00862
Record Dates: First submitted 2022-02-20; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- intermittent compression-decompression with glides (Experimental): Patients in this group will be given only intermittent compression and decompression with glides. Traction (decompression applied at knee joint with anteroposterior glide followed by compression for about 6 minutes (30 glides, 10 seconds compression and vice versa), for the duration of 4 weeks (3 days a week, alternate days)
  Interventions: Other: intermittent compression-decompression with glides
- Conventional Physical Therapy (Experimental): In this group conventional therapy will be given according to below mentioned protocol for 4 weeks (3 days a week, alternate days).
  * Hot pack /TENS for 10 minutes
  * Stretching: Hamstring(10x) and calf (10x)
  * Strengthening of periarticular muscles especially the quadriceps (straight leg raising, pillow squeeze-isometric and dynamic)
  Interventions: Other: Conventional Physical Therapy
- conventional physical therapy and intermittent compression-decompression with glides (Experimental): Patients in this group will receive the combination of conventional physical therapy andintermittent compression and decompression with glides, for 4 weeks (3 days a week, alternate days).
  Interventions: Other: conventional physical therapy and intermittent compression-decompression with glides

INTERVENTIONS:
Other: intermittent compression-decompression with glides — Patients in this group will be given only intermittent compression and decompression with glides. Traction (decompression applied at knee joint with anteroposterior glide followed by compression for about 6 minutes (30 glides, 10 seconds compression and vice versa), for the duration of 4 weeks (3 days a week, alternate days)
  Arms: intermittent compression-decompression with glides
Other: Conventional Physical Therapy — In this group conventional therapy will be given according to below mentioned protocol for 4 weeks (3 days a week, alternate days).
  * Hot pack /TENS for 10 minutes
  * Stretching: Hamstring(10x) and calf (10x)
  * Strengthening of periarticular muscles especially the quadriceps (straight leg raising, pillow squeeze-isometric and dynamic)
  Arms: Conventional Physical Therapy
Other: conventional physical therapy and intermittent compression-decompression with glides — Patients in this group will receive the combination of conventional physical therapy and intermittent compression and decompression with glides, for 4 weeks (3 days a week, alternate days).
  Arms: conventional physical therapy and intermittent compression-decompression with glides

SUMMARY:
the aim of this study is to compare the effects of intermittent compression decompression with glides with conventional physical therapy in patients having knee osteoarthritis. there are three groups in which patient will be allocated randomly. group A will receive treatment technique intermittent compression decompression with glides only while group B will be treated with conventional physical therapy protocol whereas group c patients will receive combination of intermittent compression decompression with glides along with conventional physical therapy protocol. Pre and post treatment data will be collected by using questionnaires WOMAC and KOOS. treatment will be given 3 times a week for 4 weeks.

DETAILED DESCRIPTION:
Most prevalent musculoskeletal age-related disorder worldwide is Osteoarthritis whose prevalence is supposed to rise in elderly population as it ages. knee pain is common issue contributing to OA in older population increasing with the increase of risk factor obesity and as population ages. People with Knee OA experience reduced movement, frequent chronic pain along with strength and balance compromising and face limitations in daily activities. Radio graphs of patients with knee OA show changes in lateral and medical tibiofemoral joints along with patellofemoral joint. Currently, 40% people aged above 75 years are affected with knee OA. In US, 28% adults older than 45 years of age and 37% older than 65 years of age are affected with knee OA. Knee osteoarthritis is a major age-related health problem and is leading cause of pain and disability in people.

Radiographic evidence of osteoarthritis is present in the majority of people over age 65; 80% of those over 75, Approximately 11% of those over 65 have symptomatic osteoarthritis of the knee Current guidelines recommend nonpharmacologic methods, such as physical therapy, as first-line options in the management of OA. Currently there is no medically effective treatment available. NSAIDS and acetaminophens are widely used to treat this but sometimes they fail to relieve symptoms leading to more adverse effects. Physical therapy is considered as an essential element in alleviating pain and improving physical functioning, but the data is limited. Exercise has showed improvement is walking speed, strength, functions self-efficacy along with pain alleviation during activities and enables to reduce limitation of daily. It is an urgent need to identify new effective treatment and techniques for patients with Knee OA as it is urgent health and clinical priority. Physiotherapy interventions commonly prescribed for the knee OA management includes electrotherapy along with knee isometric exercises but these are not as effective as in OA cartilage damages to as extent along with limited blood flow and reduced metabolic activity. These interventions are not enough to promote healing response of cartilage. Is supposed to promote osteoblastic activity, thus improving symptoms along with delaying the degeneration process Intermittent compression and decompression with glides has significant results in improving symptoms associated with knee OA along with betterment of quality of life. This technique is believed to delay and prevent surgical interventions as well as is cost effective treatment for patients suffering from knee OA.

Mobilization of knee joint includes the mobilization of tibiofemoral joint. This includes anterior and posterior glides with compression and decompression. Mobilization is a passive procedure performed to improve pain, increase range of motion and increase functional capability of patient, because optimal stimulus for the regeneration of the joint cartilage is intermittent compression and decompression with gliding. Manual physical therapy has also been reported to inhibit and modulate pain, induce a controlled inflammatory response that initiates healing and influences processing of pain, and alter acute inflammation in response to exercise. These could all contribute to decreased pain from muscle contract ion, improving tolerance for exercise. Joint mobilizations also modulate proprioceptive input to joint structures, prime the joint and surrounding muscles for optimal response to strengthening programs, improve muscle control and reaction times. Intermittent compression and decompression along with gliding of articular cartilage during moderate exercise activities allows synovial fluid to nourish the joint and remove waste products. This movement can also lead to thickening and increased resilience in the cartilage. Exercise also leads to increased muscle and ligamentous strength that provides stability to the joint.

Damaged articular cartilage has less healing capacity due to its low metabolic activity and limited blood circulation which permit limited response to injury. This cartilage lesion is sometime very progressive. Therefore, its early intervention is aimed to limit this progressive lesion to articular cartilage which is may be critical for decreasing the disability and chronic pain associated with osteoarthritis .Compressive forces applied on the knee joint pushes the fluid out of cartilage and during decompression it is reabsorbed, this phenomenon helps in the regeneration of cartilage by means of supplying nutrients and oxygen. Physical therapy interventions included are electrotherapy along with knee isometric exercises for management of osteoarthritis. But these interventions are not so effective and do not help in regeneration of the cartilage. Intermittent compression and decompression with glide helps to activate osteoblastic activity and improve the symptoms of osteoarthritis thus delaying the process of degeneration. The study is concerned with finding the effects of intermittent compression and decompression with glides for the knee osteoarthritis .Treatment technique in this research will substantially help to improve all the important outcomes as per literature evident .i.e. pain, disability, range of motion in patients with knee osteoarthritis. It will add innovative intervention to existing literature which will be helpful in improving quality of life in patients with knee OA.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnose with osteoarthritis of knee joint
* Age: above 40, below70 years
* Both gender (male and female) included
* Subjects with unilateral or bilateral involvement of knee
* Patients who will be able to comprehend commands.

Exclusion Criteria:

* Subject who undergone any lower limb surgery
* Subject with inflammatory joint disease of lower limb neurological disorder (motor or sensory loss).
* Intra-articular corticosteroids or hyaluronic injection during past six months.
* Subject giving history of hypersensitive skin, allergy or any other skin conditions
* Subjects with any deformity like genu varum/ genu valgum

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-10-18 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 4th week
  changes from baseline numeric pain rating scale, The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable") were taken
Knee Injury and Osteoarthritis Outcome Score (KOOS) | 4th week
  changes from baseline, The KOOS is self-administered and assesses five outcomes: pain, symptoms, activities of daily living, sport and recreation function, and knee-related quality of life were taken
Western Ontario And McMaster Osteoarthritis Index (WOMAC) | 4th week
  changes from baseline Western Ontario And McMaster Osteoarthritis Index (WOMAC) were taken. The WOMAC consists of 24 items: 5 pain, 2 stiffness, and 17 physical function items. It produces three subscale scores (pain, stiffness, and physical function) and a total score.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Affan Iqbal, PhD*, Principal Investigator — Riphah International University
Locations (4):
- Pakistan (4):
  - Chaudhary Medical Center, Haripur, Khyber Pakhtunkhwa
  - DHQ Haripur, Haripur, Khyber Pakhtunkhwa
  - Yahya Welfare Complex Hospital, Haripur, Khyber Pakhtunkhwa
  - Akhtar jahan medical center, Wah, Punjab Province

IPD SHARING:
Plan to Share IPD: No